CLINICAL TRIAL: NCT04381741
Title: CD19 CAR-T Expressing IL7 and CCL19 Combined With PD1 mAb for Relapsed or Refractory Diffuse Large B Cell Lymphoma
Acronym: CICPD
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IR2020001132
Record Dates: First submitted 2020-05-06; First posted 2020-05-11 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: diffuse large B-cell lymphoma; Chimeric antigen receptor T cell; PD1 monoclonal antibody
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD19-7×19 CAR-T plus PD1 monoclonal antibody (Experimental)
  Interventions: Biological: CD19-7×19 CAR-T plus PD1 monoclonal antibody

INTERVENTIONS:
Biological: CD19-7×19 CAR-T plus PD1 monoclonal antibody — Three different doses of CD19-7×19 CAR-T (1×106/kg、2×106/kg、3×106/kg) plus 200mg Tislelizumab every 3 weeks for 6 times

SUMMARY:
Diffuse large B-cell lymphoma (DLBCL) is the most common non-Hodgkin's lymphoma, accounting for 35% of lymphoma. Chimeric antigen receptor T cell (CAR-T) therapy is a new method to treat DLBCL. KTE-C19, published in the New England Medical Journal in December 2017, was used to treat relapsed and refractory B-cell lymphoma. One year of treatment for 111 patients, the total response rate was 82%, and the complete remission rate was 54%. However, a large number of clinical studies have shown that about 20% of patients with B-ALL and 50% of patients with B-NHL cannot achieve complete remission (CR) after CD19-CAR-T treatment. Targeting tumor microenvironment is an important new method to overcome the drug resistance of CAR-T cells. In this study, IL-7 and CCL19 were connected on the basis of traditional second generation CD19 CAR-T cells to construct novel fourth generation CAR-T cells, which can promote the infiltration, accumulation and survival of CAR-T cells in lymphoma tissue, and further enhance the anti-tumor effect of traditional CAR-T cells. At the same time, combined with four generations of CAR-T cells and PD1 monoclonal antibody, PD1 / PDL1 signal pathway was blocked, anti-tumor effect of CAR-T was improved, and immune response and long-term remission rate of DLBCL were improved.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age ≥ 18, upper limit 75, unlimited for men and women;

  (2) ECOG score 0-3;

  (3) Histologically confirmed diffuse large B-cell lymphoma (DLBCL) [according to who 2008];

  (4) CD19 was positive (immunohistochemistry or flow cytometry).

  (5) The definition of refractory or relapse of DLBCL is: no complete remission after 2-line treatment; disease progression in any treatment process, or disease stabilization time equal to or less than 6 months; or disease progression or relapse within 12 months after hematopoietic stem cell transplantation;

  (6) The previous treatment of diffuse large B cell lymphoma must include rituximab (CD20 mAb) and anthracycline;

  (7) There should be at least one measurable focus. It is required that any length of lymph node focus should be greater than 1.5cm or any length of extranodal focus should be greater than 1.0cm. PET-CT scan focuses should have uptake (SUV is greater than liver blood pool);

  (8) The absolute value of neutrophils in peripheral blood ≥ 1000 / μ L, platelet ≥ 45000 / μ L;

  (9) Heart, liver and kidney function: creatinine < 1.5mg/dl; ALT (alanine aminotransferase) / AST (aspartate aminotransferase) 2.5 times lower than the normal upper limit; total bilirubin < 1.5mg/dl; heart ejection fraction (EF) ≥ 50%;

  (10) Sufficient understanding ability and voluntary signing of informed consent;

  (11) Those with fertility must be willing to use contraceptive methods;

  (12) According to the judgment of the researchers, the expected survival time is more than 4 months;

  (13) Willing to follow visit schedule, administration plan, laboratory inspection and other test steps.

Exclusion Criteria:

* (1) History of other tumors;

  (2) Hematopoietic stem cell transplantation was performed within 6 weeks;

  (3) Any target car-t treatment was performed within 3 months before the car-t treatment;

  (4) Previous use of any commercially available PD-1 mAb;

  (5) Cytotoxic drugs, glucocorticoids and other targeted drugs were received within 2 weeks before cell collection;

  (6) Active autoimmune diseases;

  (7) Uncontrollable infection of active bacteria and fungi;

  (8) HIV infection, syphilis infection; active hepatitis B or C: hepatitis B: HBV-DNA ≥ 1000IU / ml; hepatitis C: HCV RNA positive and liver function abnormal.

  (9) Known central nervous system lymphoma.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-06-18 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 3 months
  Objective response rate of the combination of CD19 CAR-T Expressing IL7 and CCL19 and PD1 mAb

SECONDARY OUTCOMES:
progression-free survival | 2 years
  progression-free survival of the combination of CD19 CAR-T Expressing IL7 and CCL19 and PD1 mAb
overall survival | 2 years
  overall survival of the combination of CD19 CAR-T Expressing IL7 and CCL19 and PD1 mAb
Duration of Overall Response | 2 years
  Duration of Overall Response of the combination of CD19 CAR-T Expressing IL7 and CCL19 and PD1 mAb
Relapse rate | 2 years
  Relapse rate of the combination of CD19 CAR-T Expressing IL7 and CCL19 and PD1 mAb

CONTACTS AND LOCATIONS:
Overall Officials: Wenbin Qian, MD, PhD, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-20): https://cdn.clinicaltrials.gov/large-docs/41/NCT04381741/Prot_SAP_000.pdf
  • Informed Consent Form (2020-03-20): https://cdn.clinicaltrials.gov/large-docs/41/NCT04381741/ICF_001.pdf